CLINICAL TRIAL: NCT03567213
Title: Investigation on the Cortical Communication (CortiCom) System
Acronym: CortiCom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00167247; UH3NS114439 (NIH)
Record Dates: First submitted 2018-05-21; First posted 2018-06-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Tetraplegia; Locked-in Syndrome; Brainstem Stroke; Amyotrophic Lateral Sclerosis
Keywords: Tetraplegia; ALS; Locked-in Syndrome; Brainstem stroke; Brain Computer Interface; Rehabilitation; Stroke; Hopkins
MeSH Terms: conditions — Quadriplegia; Locked-In Syndrome; Brain Stem Infarctions; Amyotrophic Lateral Sclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Surgical implantation of the CortiCom system (Experimental)
  Interventions: Device: Surgical implantation of CortiCom system

INTERVENTIONS:
Device: Surgical implantation of CortiCom system — Implantation of Cortical communication system, consisting of one or two Electrocorticography (ECoG) grids connected to a transcutaneous patient pedestal.

SUMMARY:
The CortiCom system consists of 510(k)-cleared components: platinum PMT subdural cortical electrode grids, a Blackrock Microsystems patient pedestal, and an external NeuroPort Neural Signal Processor. Up to two grids will be implanted in the brain, for a total channel count of up to 128 channels, for six months. In each participant, the grid(s) will be implanted over areas of cortex that encode speech and upper extremity movement.

DETAILED DESCRIPTION:
The successful adoption of brain-computer interfaces (BCIs) as assistive technologies (ATs) for disabled populations depends on the ability to elicit rapid, intuitive, and reliable control signals. To date, it is not known which sources of neural information provide the most natural and efficient means of control. This study will directly assess the efficacy of two sources of neural control signals, speech and motor cortex, for BCI control of software and devices using investigators' Cortical Communication (CortiCom) system.

The CortiCom system consists of 510(k)-cleared components: platinum PMT subdural cortical electrode grids, a Blackrock Microsystems patient pedestal, and an external NeuroPort Neural Signal Processor. Up to two grids will be implanted in the brain, for a total channel count of up to 128 channels, for six months. In each participant, the grid(s) will be implanted over areas of cortex that encode speech and upper extremity movement.

Investigators' study will be the first to investigate the efficiency and intuitiveness of two contrasting neural control strategies for BCI: Motor imagery and speech. As the first study to chronically and simultaneously record from human speech and motor regions, this study seeks to achieve the following:

* demonstrate the ability to decode intended upper extremity movements using information decoded from primary motor cortex arm/hand area;
* demonstrate the ability to decode intended speech from articulatory speech cortex; and
* determine the most effective and intuitive user strategies (e.g. imagined speech or imagined movement) and optimal neural sources for brain-computer interactions,

The patient populations targeted in this study are amyotrophic lateral sclerosis (ALS), brainstem stroke, locked-in syndrome (LIS), and tetraplegia. Individuals within these populations may have normal cortical function and cognition while suffering from motor or combined speech and motor deficits.

Based on research by colleagues, as well as investigators' own experience working with participants affected by epilepsy implanted with high density electrocorticographic grids, investigators hypothesize that long-term recording of neural activity from the targeted cortical areas may provide a new communication channel for these clinical populations. The utilization of high-channel-count (up to 128 channel) ECoG grids, in combination with simultaneous coverage of speech and motor cortex, will enable investigations into the performance of speech-mediated and motor-mediated control efficacy as applied to a variety of end effectors, such as computers, tablets, headsets for virtual or augmented reality, smart lights, televisions, and assistive technologies. Additionally, eye-tracking may be utilized in combination with neural commands to improve target selection performance and ease.

Through this study, investigators will assess the performance of speech- and motor-mediated control using chronic, high-channel count ECoG grid neural implants in pursuit of a high-performing, clinically beneficial BCI assistive technology.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of tetraplegia (quadriplegia), brainstem stroke , amyotrophic lateral sclerosis (ALS) or Locked-in Syndrome (LIS)
* Tetraplegia diagnosis, ALS diagnosis, stroke, or LIS etiology onset occurred at least one year prior to enrollment
* Complete or incomplete tetraplegia (quadriplegia), tetraparesis (quadriparesis), or severe ataxia. In addition, these motor impairments may be combined with severe motor-related speech impairment (dysarthria or anarthria), as in LIS.
* 22-70 years
* Meeting surgical safety criteria, including surgical clearance by the participant's primary healthcare provider, study physicians, and any necessary consultants
* Ability to communicate reliably, such as through eye movement
* Willingness and ability to provide informed consent
* Screened by rehabilitation psychologist with a result showing that the participant has a stable psychosocial support system with caregiver capable of monitoring participant throughout the study
* Ability and willingness to travel up to 100 miles to study location up to three days per week for the duration of the study
* Ability to understand and comply with study session instructions
* Participant consents to the study and still wishes to participate at the time of the study

Exclusion Criteria:

* Performance on formal neuropsychological testing that indicates significant psychiatric conditions or cognitive impairments that would interfere with obtaining informed consent or fully participating in study activities.
* Suicide attempt or persistent suicidal ideation within the past 12 months.
* Implanted devices that are incompatible with MRI, which may include pacemakers, cardiac defibrillators, spinal cord or vagal nerve stimulators, deep brain stimulators, and cochlear implants.
* History of substance abuse, narcotic dependence, or alcohol dependence in past 24 months
* Medical conditions contraindicating surgery of a chronically implanted device (e.g. osteomyelitis, diabetes, hepatitis, any autoimmune disease/disorder, epilepsy, skin disorders causing excessive skin sloughing or poor wound healing, blood or cardiac disorder requiring chronic anti-coagulation)
* Other chronic, unstable medical conditions that could interfere with subject participation.
* Presence of pre-surgical findings in anatomical, functional, and/or vascular neuroimaging that makes achieving implant locations within desired risk levels too challenging (to be decided by neurological and neurosurgical team)
* Prior cranioplasty
* Inability to undergo MRI or anticipated need for an MRI during the study period
* Participants with active infections or unexplained fever
* Participants with other morbid conditions making the implantation of the recording elements unsafe; not limited to: significant pulmonary, cardiovascular, metabolic, or renal impairments making the surgical procedure unsafe
* Pregnancy (confirmation through blood test)
* Nursing an infant, planning to become pregnant, or not using adequate birth control
* Corrected vision poorer than 20/100
* HIV or AIDS infection
* Existing scalp lesions or skin breakdown
* Chronic oral or intravenous use of steroids or immunosuppressive therapy
* Active cancer within the past year or requires chemotherapy
* Uncontrolled autonomic dysreflexia within the past 3 months
* Hydrocephalus with or without an implanted ventricular shunt
* Participants in whom it is medically contraindicated to stop anti-coagulant medications during surgery

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to device explantation | 26 weeks
  This study outcome will be considered successful if the device is not explanted during the 26-week period of the study. Explantation of the device prior to the completion of the 26-week period implies that the device is putting the subject at risk (e.g. through a serious infection at the implantation site) and therefore must be removed.

SECONDARY OUTCOMES:
Success rate in controlling the brain computer interface, i.e. ratio of successful trials to total trials. | 26 weeks
  One or more participants demonstrates successful use of the CortiCom system in which motor and/or speech neural signals can be decoded to provide control signals for software and devices. Efficacy is assessed in terms of accuracy, i.e. how often the participant is able to select a desired target.
Speed of brain-computer interface control, i.e. time to complete successful trials (in seconds). | 26 weeks
  One or more participants demonstrates successful use of the CortiCom system in which motor and/or speech neural signals can be decoded to provide control signals for software and devices. Efficacy is therefore also assessed in terms of how long it takes to select the target.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan E Crone, MD, Principal Investigator — Professor of Neurology
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD from published results will be made available upon reasonable request to corresponding authors and/or will be uploaded to a data archive for the BRAIN Initiative in compliance with its data sharing consortium.
Supporting Information: Analytic Code
Time Frame: IPD and associated analytic code will be made available upon publication of research results and will remain available for the duration of the funded project.

REFERENCES:
- [Derived] Candrea DN, Angrick M, Luo S, Ganji R, Coogan C, Milsap GW, Rosenblatt KR, Uchil A, Clawson L, Maragakis NJ, Vansteensel MJ, Tenore FV, Ramsey NF, Fifer MS, Crone NE. Longitudinal study of gesture decoding in a clinical trial participant with ALS. medRxiv [Preprint]. 2025 Oct 3:2025.09.26.25335804. doi: 10.1101/2025.09.26.25335804. PMID 41256173
- [Derived] Angrick M, Luo S, Rabbani Q, Joshi S, Candrea DN, Milsap GW, Gordon CR, Rosenblatt K, Clawson L, Maragakis N, Tenore FV, Fifer MS, Ramsey NF, Crone NE. Real-time detection of spoken speech from unlabeled ECoG signals: a pilot study with an ALS participant. J Neural Eng. 2025 Oct 6;22(5):056023. doi: 10.1088/1741-2552/ae0965. PMID 40972658
- [Derived] Candrea DN, Shah S, Luo S, Angrick M, Rabbani Q, Coogan C, Milsap GW, Nathan KC, Wester BA, Anderson WS, Rosenblatt KR, Uchil A, Clawson L, Maragakis NJ, Vansteensel MJ, Tenore FV, Ramsey NF, Fifer MS, Crone NE. A click-based electrocorticographic brain-computer interface enables long-term high-performance switch scan spelling. Commun Med (Lond). 2024 Oct 22;4(1):207. doi: 10.1038/s43856-024-00635-3. PMID 39433597
- [Derived] Angrick M, Luo S, Rabbani Q, Joshi S, Candrea DN, Milsap GW, Gordon CR, Rosenblatt K, Clawson L, Maragakis N, Tenore FV, Fifer MS, Ramsey NF, Crone NE. Real-time detection of spoken speech from unlabeled ECoG signals: A pilot study with an ALS participant. medRxiv [Preprint]. 2024 Sep 22:2024.09.18.24313755. doi: 10.1101/2024.09.18.24313755. PMID 39371161
- [Derived] Wyse-Sookoo K, Luo S, Candrea D, Schippers A, Tippett DC, Wester B, Fifer M, Vansteensel MJ, Ramsey NF, Crone NE. Stability of ECoG high gamma signals during speech and implications for a speech BCI system in an individual with ALS: a year-long longitudinal study. J Neural Eng. 2024 Jul 12;21(4):10.1088/1741-2552/ad5c02. doi: 10.1088/1741-2552/ad5c02. PMID 38925110
- [Derived] Angrick M, Luo S, Rabbani Q, Candrea DN, Shah S, Milsap GW, Anderson WS, Gordon CR, Rosenblatt KR, Clawson L, Tippett DC, Maragakis N, Tenore FV, Fifer MS, Hermansky H, Ramsey NF, Crone NE. Online speech synthesis using a chronically implanted brain-computer interface in an individual with ALS. Sci Rep. 2024 Apr 26;14(1):9617. doi: 10.1038/s41598-024-60277-2. PMID 38671062
- [Derived] Crone N, Candrea D, Shah S, Luo S, Angrick M, Rabbani Q, Coogan C, Milsap G, Nathan K, Wester B, Anderson W, Rosenblatt K, Clawson L, Maragakis N, Vansteensel M, Tenore F, Ramsey N, Fifer M, Uchil A. A click-based electrocorticographic brain-computer interface enables long-term high-performance switch-scan spelling. Res Sq [Preprint]. 2023 Sep 25:rs.3.rs-3158792. doi: 10.21203/rs.3.rs-3158792/v1. PMID 37841873
- [Derived] Angrick M, Luo S, Rabbani Q, Candrea DN, Shah S, Milsap GW, Anderson WS, Gordon CR, Rosenblatt KR, Clawson L, Maragakis N, Tenore FV, Fifer MS, Hermansky H, Ramsey NF, Crone NE. Online speech synthesis using a chronically implanted brain-computer interface in an individual with ALS. medRxiv [Preprint]. 2023 Jul 1:2023.06.30.23291352. doi: 10.1101/2023.06.30.23291352. PMID 37425721
- See also: Additional study information — https://www.hopkinsmedicine.org/neurology_neurosurgery/clinical-trials/brain-computer-interface.html